CLINICAL TRIAL: NCT02105740
Title: Hypnosis as a Complementary Practice in Pain Management, Anxiety and Depression in Oncological Patients
Brief Title: Hypnosis in Pain Management, Anxiety and Depression in Oncological Patients
Acronym: HPMADOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gil Montenegro (Other)
Collaborators: University of Brasilia (Other)
Responsible Party: Sponsor-Investigator, Gil Montenegro, PhD student in medical science, University of Brasilia
Organization: University of Brasilia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UNB19739513900000030
Record Dates: First submitted 2014-03-27; First posted 2014-04-07 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Pain; Depression Anxiety Disorder
Keywords: BEHAVIORAL; HYPNOSIS; ANXIETY; DEPRESSION
MeSH Terms: conditions — Pain; Behavior; Anxiety Disorders; Depression | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnosis (Experimental): Use of hypnosis in the reduction of the levels of pain, depression and anxiety.
  Interventions: Behavioral: Hypnosis
- Control (Active Comparator): Comparison of the effects of hypnosis between the control group and the experimental group regarding pain, anxiety and depression with the application of the scales.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Hypnosis — The hypnosis intervention consists of two 40-minute sessions, with an interval of 7 days between them, emphasizing the pain blocking, the well-being of the patient and the reduction of the symptoms of anxiety and depression of the same.
  Arms: Hypnosis
Behavioral: Control — The control and experimental groups respond in 3 different moments to Visual Analogue Scale (VAS) for the evaluation of pain, and to Hospital Anxiety and Depression Scale (HADS) to evaluate depression and the anxiety. The first meeting will be made before the hypnosis. In the second meeting, within an interval of 7 days, the scales will be applied in all patients. Before applying the scales, the hypnosis group will be submitted to the session. The third meeting will occur two weeks later, where the scales will be only applied to compare the groups.
  Arms: Control

SUMMARY:
The aim of this trial is to compare and evaluate the effects of hypnosis in cancer patients, to reduce the level of pain, anxiety and depression. The comparison was made through the scores on the Visual Analogue Scale (VAS) and the Hospital Anxiety and Depression Scale (HADS).

DETAILED DESCRIPTION:
Volunteers cancer patients of both gender, aged between 40 and 70 years, susceptible to hypnosis, with pain scores ≥ 3 measured by Visual Analogue Scale (VAS), will be randomized into two groups of 12 participants each. They might or might not present metastasis, whether or not performed cancer surgery, regardless of the location of the primary tumor, with or without concomitant surgical indication. It will be used the Visual Analogue Scale (VAS) and Hospital Anxiety and Depression Scale (HADS) at 3 different times: at baseline, after 7 days and after 2 weeks of the first assessment. It will be done, in the hypnosis group, an hypnosis intervention. It consists of two 40-minute sessions, with an interval of 7 days between them, emphasizing the pain blocking, the well-being of the patient and the reduction of the symptoms of anxiety and depression. Then, it will be evaluated the intensity of the pain as well as depression and anxiety in both groups. Finally, the results of both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Both sexes
* Aged 40-70 years susceptible to hypnosis
* Who have cancer of the digestive tract and pain resulting from this cancer treatment These may or may not have metastasis, have done or not cancer surgery, regardless of the location of the primary tumor or its presence,with or without concomitant surgical indication.This will include patients who have pain scores ≥ 3 in the Visual Analogue Scale (VAS).

Exclusion Criteria:

* Patient not suggestible to hypnosis
* Psychotropic drug users,
* Patients with severe psychiatric disorder, except depression and anxiety

  ,- Patient terminally ill cancer
* Patients with tumor or cancer metastasis in the central nervous system, _ Deaf and people with mental disabilities and cognitive.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GIL MONTENEGRO, DOUTORANDO, Principal Investigator
Locations (1):
- UNB- Universidade de Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardia A, Barton DL, Prokop LJ, Bauer BA, Moynihan TJ. Efficacy of complementary and alternative medicine therapies in relieving cancer pain: a systematic review. J Clin Oncol. 2006 Dec 1;24(34):5457-64. doi: 10.1200/JCO.2006.08.3725. PMID 17135649
- [Background] Lalla RV, Sonis ST, Peterson DE. Management of oral mucositis in patients who have cancer. Dent Clin North Am. 2008 Jan;52(1):61-77, viii. doi: 10.1016/j.cden.2007.10.002. PMID 18154865
- [Background] Montgomery GH, Bovbjerg DH, Schnur JB, David D, Goldfarb A, Weltz CR, Schechter C, Graff-Zivin J, Tatrow K, Price DD, Silverstein JH. A randomized clinical trial of a brief hypnosis intervention to control side effects in breast surgery patients. J Natl Cancer Inst. 2007 Sep 5;99(17):1304-12. doi: 10.1093/jnci/djm106. Epub 2007 Aug 28. PMID 17728216
- [Background] Porter LS, Keefe FJ. Psychosocial issues in cancer pain. Curr Pain Headache Rep. 2011 Aug;15(4):263-70. doi: 10.1007/s11916-011-0190-6. PMID 21400251
- [Background] Spiegel D, Bloom JR. Group therapy and hypnosis reduce metastatic breast carcinoma pain. Psychosom Med. 1983 Aug;45(4):333-9. doi: 10.1097/00006842-198308000-00007. PMID 6622622
- [Background] Trijsburg RW, van Knippenberg FC, Rijpma SE. Effects of psychological treatment on cancer patients: a critical review. Psychosom Med. 1992 Jul-Aug;54(4):489-517. doi: 10.1097/00006842-199207000-00011. PMID 1502290
- [Background] Landier W, Tse AM. Use of complementary and alternative medical interventions for the management of procedure-related pain, anxiety, and distress in pediatric oncology: an integrative review. J Pediatr Nurs. 2010 Dec;25(6):566-79. doi: 10.1016/j.pedn.2010.01.009. Epub 2010 Mar 12. PMID 21035021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process was conducted from March to December 2015. Thirty nine patients were invited. They had cancer of digestive tract from both genders, of 40-70 years, with pain scores ≥ 3 by (EVA). Were excluded: patients that used psychotropic drugs, with psychiatric disorders, terminally ill cancer, hearing impaired and mentally disabled.
Pre-assignment Details: Were excluded: 3 patients weren't suggestible, 3 patients who had terminal cancer, 2 patients who reported low scores, and 7 patients for other reasons such as religious issues or not accepting the technique. One patient dropped out the treatment because he had limited mobility to return to the hospital.
Groups:
- Hypnosis: Use of hypnosis in the reduction of the levels of pain, depression and anxiety.
  Hypnosis: The hypnosis intervention consists of two sessions of 40-minute, with an interval of 7 days between them, emphasizing the pain blocking, the well-being of the patient and the reduction of the symptoms of anxiety and depression.
- Control: Comparison of the effects of hypnosis between the control group and the hypnosis group regarding pain, anxiety and depression with the application of the scales.
  Control x Hypnosis Group: The control and hypnosis groups respond in 3 different distinct moments, with the Visual Analogue Scale (VAS) for the evaluation of pain, and the Hospital Anxiety and Depression Scale (HADS) to evaluate the depression and the anxiety. The first evaluation will be made before the research. The second within an interval of 7 days, so being that in the experimental group the same will happen after the hypnosis session and in the control group, after the follow-up visit. The third evaluation will occur two weeks later, in order to provide a follow-up to assess the efficacy of the technique. The experimental group and the control group will be compared in relation to the intensity of the pain, depression and anxiety.
Period: Overall Study
Arm/Group | Hypnosis | Control
Started | 12 (Application of EVA and HADS scales and after that application of hypnosis intervention) | 12 (Application of EVA and HADS scales)
Second | 12 (Intervention with hypnosis and application of EVA scales and HADS (n = 12)) | 11 (Application of EVA and HADS scales. One accompanying lost)
Completed | 12 (Application of EVA and HADS scales and data analysis) | 11 (Application of EVA and HADS scales and data analysis)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participated in the study, patients with cancer of the digestive tract of the Clinic Palliative Care of Brasilia Base Hospital (HBDF) who present pain ≥ 3 on the Visual Analogue Scale
Groups:
- Hypnosis: Use of hypnosis to reduct the levels of pain, depression and anxiety.
  Hypnosis: The hypnosis intervention consists of two sessions of 40-minute, with an interval of 7 days between them, emphasizing the pain blocking, the well-being of the patient and the reduction of the symptoms of anxiety and depression of the same.
- Control: Comparison of the effects of hypnosis between the control group and the experimental group regarding pain, anxiety and depression with the application of the scales.
  Control : The control and experimental groups respond in 3 different moments to Visual Analog Scale (VAS) for the evaluation of pain, and to Hospital Anxiety and Depression Scale (HADS) to evaluate depression and the anxiety. The first meeting was made before the hypnosis. In the second meeting, within an interval of 7 days, the scales were applied in all patients. Before applying the scales, the hypnosis group was submitted to the session. The third meeting occurred two weeks later, where the scales were only applied to compare the groups.
- Total: Total of all reporting groups
Arm/Group | Hypnosis | Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (6.6) | 55.8 (7.5) | 55.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 12 | 12 | 24
Pain [Mean (Standard Deviation); unit: units on a scale] — The Visual Analogue Scale (VAS) consist in a straight line in ascending order from left to right, which may be numbered from 0 to 10, in which the patient report pain intensity. Values above 03 are already considered significant for pain.
  units on a scale | 7.3 (2.4) | 5.6 (2.0) | 6.4 (2.3)
Anxiety [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS) has 14 questions, seven are aimed at evaluating anxiety (HADS-A) and seven for depression (HADS-D). Each item can be scored from 0 to 3, establish a maximum score of 21 points for each subscale. Values ≥ 9 for each subscales indicate the symptom.
  units on a scale | 11.5 (4.6) | 11.3 (4.4) | 11.4 (4.4)
Depression [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale has 14 questions, seven are aimed at evaluating anxiety (HADS-A) and seven for depression (HADS-D). Each item can be scored from zero to three, establish a maximum score of 21 points for each scale adopted as the cut points for both ≥ 9 subscales to the symptom diagnosis
  units on a scale | 9.8 (5.3) | 9.0 (3.8) | 9.4 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Score in the Visual Analogue Scale
Description: Comparison was made through the scores in the Visual Analogue Scale (VAS) to measure the effect of hypnosis in pain among the 12 patients of the hypnosis group comparing to the 11 patients of the control group. The scale ranged from 0 to 10 points, without subscales. The better outcome occurs when the mean of the second or the third week decrease 3 points comparing with the first week, or when the mean of the third week decrease 3 points comparing with the second week.
Time Frame: The study was done with each patient in the first three consecutive weeks after randomization
Population: 24 cancer patients were allocated. They were aged between 40-70 years, of both genders, with pain scores ≥ 3 measured by Visual Analogue Scale (VAS). One patient of the control group left the research.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hypnosis: Use of hypnosis to change the levels of pain.
  Hypnosis: The hypnosis intervention consists of two 40-minute sessions, with an interval of 7 days between them, emphasizing the pain blocking, the well-being of the patient and the reduction of the symptoms.
- Control: Comparison of the effects of hypnosis between the control group and the hypnosis group regarding pain with the application of the Visual Analogue Scale (VAS).
  Control x Hypnosis Group: The control and the hypnosis groups respond in 3 different distinct moments, using the Visual Analogue Scale (VAS) to evaluate the pain. The first evaluation was made before the research. The second within an interval of 7 days, so being that in the experimental group the same will happen after the hypnosis session and in the control group after the follow-up visit. The third evaluation was made two weeks later, in order to provide a follow-up to assess the efficacy of the technique.
Arm/Group | Hypnosis | Control
Number analyzed (Participants) | 12 | 11
units on a scale
  First Week | 7.33 (2.38) | 5.58 (2.06)
  Second Week | 3.67 (2.77) | 5.67 (3.36)
  Third Week | 2.08 (2.61) | 4.75 (3.13)
Statistical Analysis 1: Comparison: Hypnosis vs Control; The clinical significance was considered with a difference of 3 points on the Visual Analogue Scale (VAS) for both arms with a statistical power of 95%, significance level of 5%. Statistical analysis first compared the difference of means between hypnosis and control groups during three weeks; Test type: Superiority or Other; p = 0.034, ANOVA; Mean Difference (Final Values) = 2.67, 95% CI 2-sided [0.224 to 5.110], Standard Deviation 1.178
Statistical Analysis 2: Comparison: Hypnosis; The clinical significance was considered with a difference of 3 points on the Visual Analogue Scale (VAS) with a statistical power of 95%, significance level of 5%. Statistical analysis compared the difference in pain average between the first and the second week in the hypnosis group; Test type: Superiority or Other; p = 0.004, ANOVA; Mean Difference (Net) = 3.66, 95% CI 2-sided [1.253 to 6.080], Standard Deviation 0.856
Statistical Analysis 3: Comparison: Hypnosis; The clinical significance was considered with a difference of 3 points on the Visual Analogue Scale (VAS) with a statistical power of 95%, significance level of 5%. Statistical analysis compared the difference in pain average between the first and the third week in the hypnosis group; Test type: Superiority or Other; p = 0.000, ANOVA; Mean Difference (Net) = 5.25, 95% CI 2-sided [2.918 to 7.582], Standard Deviation 0.827

2. Secondary Outcome: Change of Anxiety and Depression in the Hospital Anxiety and Depression Scale (HADS)
Description: Comparison was made through the scores in the Hospital Anxiety and Depression Scale (HADS) to measure the effect of hypnosis in anxiety and depression among the 12 patients of the hypnosis group comparing to the 11 patients of the control group. The scale has 14 items, seven of which are directed to the evaluation of anxiety (HADS-A) and seven to depression (HADS-D). Each item can be scored from zero to three, establishing a score range of 0 to 21 points for each subscale. The better outcome occurs when the mean is lower or equal to 9 for each subscale. The subscales are independent for each result of depression and anxiety.
Time Frame: The study was done with each patient in the first three consecutive weeks after randomization
Population: Were allocated 24 cancer patients, aged between 40-70 years, of both genders, with depression and anxiety score ≥ 9 in Hospital Anxiety and Depression Scale (HADS). One patient of the control group left the research.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hypnosis: Use of hypnosis in the reduction of the levels depression and anxiety.
  Hypnosis: The hypnosis intervention consists of two 40-minute sessions, with an interval of 7 days between them, emphasizing the pain blocking, the well-being of the patient and the reduction of the symptoms of anxiety and depression of the same.
- Control: Comparison of the effects of hypnosis between the control group and the experimental group regarding anxiety and depression with the application of the Hospital Anxiety and Depression Scale (HADS).
  Control x Experimental Group: The control and experimental groups respond in 3 different distinct moments, with the Hospital Anxiety and Depression Scale (HADS) to evaluate depression and anxiety. The first evaluation was made before the research. The second within an interval of 7 days, so being that in the experimental group the same will happen after the hypnosis session and in the control group after the follow-up visit. The third evaluation was two weeks later, in order to provide a follow-up to assess the efficacy of the technique. The experimental group and the control group was compared in relation to the intensity of the depression and anxiety
Arm/Group | Hypnosis | Control
Number analyzed (Participants) | 12 | 11
units on a scale
  Anxiety First Week | 11.50 (4.60) | 11.33 (4.41)
  Anxiety Second Week | 8.17 (3.76) | 11.50 (2.43)
  Anxiety Third Week | 7.50 (3.39) | 8.89 (5.96)
  Depression First Week | 9.75 (5.32) | 9.00 (3.76)
  Depression Second Week | 7.00 (5.46) | 8.75 (4.75)
  Depression Third Week | 6.25 (3.98) | 7.75 (5.10)
Statistical Analysis 1: Comparison: Hypnosis vs Control; Statistical analysis evaluated if the difference of averages of anxiety at the hypnosis and control groups in the third week; Test type: Superiority or Other; Mean Difference (Final Values) = 1.39
Statistical Analysis 2: Comparison: Hypnosis vs Control; Statistical analysis evaluated if the difference of averages of depression at the hypnosis and control groups in the third week; Test type: Superiority or Other; Mean Difference (Final Values) = 1.5

ADVERSE EVENTS:
Groups:
- Control: Comparison of the effects of hypnosis between the control group and the experimental group regarding pain, anxiety and depression with the application of the scales.
  Control x Experimental Group: The control and experimental groups respond in 3 different distinct moments, with the Visual Analog Scale (VAS) for the evaluation of pain, and the Hospital Anxiety and Depression Scale (HADS) to evaluate the depression and the anxiety. The first evaluation will be made before the research. The second within an interval of 7 days, so being that in the experimental group the same will happen after the hypnosis session and in the control group after the follow-up visit. The third evaluation will be two weeks later, in order to provide a follow-up to assess the efficacy of the technique. The experimental group and the control group will be compared in relation to the intensity of the pain, depression and anxiety
Arm/Group | Hypnosis | Control
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
The hypnosis group were not blinded to the intervention. A short follow-up was given to each patient. The use of drugs was imbalanced among participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No